CLINICAL TRIAL: NCT05206747
Title: A Randomized Control Trial of the Effectiveness of Blue-blocking Glasses for Mania in Inpatients With Bipolar Disorder
Brief Title: Ottawa Sunglasses at Night for Mania Study
Acronym: OSAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20210790-01H
Record Dates: First submitted 2022-01-07; First posted 2022-01-25 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Mania; Sleep; Bipolar Disorder
Keywords: Blue Blocking Glasses; Randomized
MeSH Terms: conditions — Mania; Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: The investigators plan to conduct an up to two-week single-blind, randomized controlled trial of blue-blocking glasses added to treatment as usual for mania. Participants will be randomized 1:1 to wearing blue blocking glasses or lightly-tinted glasses. To ensure temporal and geographic balance, randomization will be stratified by the three sites in blocks of four.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will be informed that the investigators are studying the effects of two different types of light filters without more detail so they will not know which is the experimental vs. control condition. With possible un-blinding from other sources of information and lens color, the investigators will assess the integrity of the blind by asking participants whether they thought they received the experimental or the control glasses at the end of the study. Participates will also be encouraged not to share details of their glasses assignment with other participants and physicians to avoid unblinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blue-blocking glasses (Experimental): Participants will wear orange/amber colored lenses that filter wavelengths of light in the blue spectrum while awake from 6 p.m. to 8 a.m.
  Interventions: Device: Blue-blocking glasses
- Lightly-tinted glasses (Sham Comparator): This control will involve glasses that selectively filter short wavelength (e.g., ultraviolet), but not visible blue light during the same time window. Participants will wear these glasses while awake from 6 p.m. to 8 a.m.
  Interventions: Device: Lightly-tinted glasses

INTERVENTIONS:
Device: Blue-blocking glasses — It will transmit 45% of visible light with the following light transmission profile.
  Arms: Blue-blocking glasses
Device: Lightly-tinted glasses — It will also filter short wavelength light but at a lower threshold with near identical transmission above this threshold. It will transmit 91% of visible light with the following light transmission profile.
  Arms: Lightly-tinted glasses

SUMMARY:
Mania is a serious condition. Symptoms of mania include decreased sleep, increased energy, changes in mood, thinking, and behavior. Dark therapy, which involves placing patients in a dark room for 14 hours overnight, can effectively treat mania, but is not practical. Dark therapy is also unpleasant. However, similar effects on the brain can be created from blocking only blue light with glasses. This preserves the wearer's ability to see and move safely. A trial of blue-blocking glasses for mania in Norway produced dramatic improvements in manic symptoms within three days of hospitalization. Mania both disrupts the sleep-wake cycle and is triggered by short and interrupted sleep. Examples of triggers include shift work and travel across time zones. Therefore, mania involves the "day-night" clock in the brain. The rhythm of the brain's clock is set by special sensors in the eye that identify daytime from blue light. If light does not include this blue spectrum, this informs the brain it is nighttime. In spite of the obvious potential of blue blocking glasses for mania, there has been no confirmatory study of this simple treatment in the five years since the initial Norwegian trial. Without a second study, this treatment will not find its way into routine clinical care. The investigators will conduct a randomized controlled trial of blue-blocking glasses for mania in hospitalized patients. The investigators will also assess activity, sleep, and saliva melatonin (a hormone secreted in the brain at night) to see how this treatment works. If our trial confirms that blue-blocking glasses are effective, this treatment could help those suffering with mania return to their life more quickly. Medications for mania can also cause serious side-effects and having glasses as a treatment option might also reduce the amount of medicine needed to get well. Blue-blocking glasses could be a low-cost non-medication treatment. The investigators will look at how they could put this treatment into practice as part of everyday care.

DETAILED DESCRIPTION:
The purpose of this research project is to determine the effectiveness of blue-blocking glasses as adjunctive treatment for mania in bipolar disorder, assess circadian mechanisms, and provide information to improve translation to real-world practice settings. The investigators propose to conduct a confirmatory and more definitive clinical trial of blue-blocking glasses for mania and explore the putative role of circadian factors in mechanisms of action.

The primary objective is to specifically determine whether blue-blocking glasses are effective at reducing manic symptoms in inpatients beyond any general reduction in light exposure. This represents an advance on prior study, which compared them to clear lenses. For reasons outlined in the background, the investigators hypothesis that adding blue-blocking glasses to pharmacological treatment as usual for mania will improve symptoms, as measured by the clinician administered rating scales.

The secondary objectives relate to understanding how the reduction in manic symptoms with blue blocking glasses corresponds to changes in circadian rhythms. Not all patient with mania will be able to participate in this portion of the protocol (relevant to Aim 2 below) and it will subsequently be performed in a subset of patients, who are both capable and interested in adhering to the protocol, and at sites able to implement. At this time, the investigators anticipate this portion of the protocol being administered at the two campuses of The Ottawa Hospital. The investigators hypothesize that changes in circadian rhythms will be correlated to improvement in manic symptoms and thus a likely mechanisms of action.

The investigators also plan to conduct qualitative interviews to inform future implementation of this or related interventions (Aim 3).

Aim 1 (Effectiveness): To compare the effectiveness (change in Young Mania Rating Scale) of blue-blocking glasses to lightly tinted glasses as an adjunctive therapy with treatment as usual for psychiatric inpatients with mania.

Aim 2 (Support of Mechanism): To assess whether the reduction in manic symptoms with blue blocking glasses relates to the degree of changes in circadian rhythms (based on melatonin release curves, body temperature, heart rate, and the rest-activity cycle derived from actigraphy) and sleep (subjective and based on actigraphy).

Aim 3 (Translation to Practice): To improve translation to real-world practice settings, qualitative interviews with staff and patients will be performed using the Reach Effectiveness Adoption Implementation (RE-AIM) model.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 to 70 years of age
* Have a Diagnostic and Statistical Manual of Mental Disorders (5th Edition) defined manic symptoms that persist beyond the physiological effects of a substance
* Be willing to have investigators obtain information from the treatment team and electronic medical record
* Participants must be able to read and understand English or French.
* Be willing and able to provide informed consent.
* (Sub-study only): Meet the safety specifications for the devices in the sub-study, according to their user manuals

Exclusion Criteria:

* Have severe eye disease or trauma
* Have a history of traumatic brain injury.
* Have sleep apnea
* (Sub-study only): Have current exogenous melatonin intake

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Change in the Young Mania Rating Scale | Baseline to Week 2 (End of Study)
  The Young Mania Rating Scale is used to evaluate the severity of manic symptoms at baseline and over time in individuals with mania. It is an 11-item scale and total score ranges from 0 to 60 where higher scores indicate more severe mania, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in manic symptoms. Total score ≤12 indicates remission (13-19=minimal symptoms; 20-25=mild mania, 26-37=moderate mania, 38-60=severe mania). We will model differences between groups in the primary outcome using linear mixed models (group by time interaction) including a random intercept term for participant.

SECONDARY OUTCOMES:
Amount of antipsychotic (in chlorpromazine equivalents) and benzodiazepine used (in lorazepam equivalents) | Baseline to Week Two (End of Study)
  Medication use will be abstracted from the medication administration record to assess need for scheduled and as needed antipsychotics and benzodiazepines.
Total number of medications needed | Baseline to Week Two (End of Study)
  Medication use will be abstracted from Medication Administration Records of the Electronic Medical Record.
Differences in sleep efficiency as estimated from actigraphy | Baseline to Two Weeks (End of Study)
  In a subsample of the study, validated monitors will also be used for non-invasive and wireless continuous monitoring of movements through wrist actigraphy (Actiwatch Spectrum Plus, Philips Healthcare, Bend, USA)
Change in the Patient Mania Questionnaire - 9-Item Scale for Assessing and Monitoring Manic Symptoms (PMQ-9) | Baseline; Week One; Two Week (End of Study)
  All items in the Patient Mania Questionnaire included time frame and stem-phrase format of "Over the past week, how often have you….". The Patient Mania Questionnaire item responses ranged from 0 to 3 with 0 indicating "not at all," 1 indicating "several days," 2 indicating "more than half of days," and 3 indicating "nearly every day." Item scores were added so that the total score ranged from 0 to 27 with higher scores representing greater severity.
Change in the Digital Self-Report Survey of Mood for Bipolar Disorder - 6-Item Digital Survey Measuring Mood Changes in Bipolar Disorder (digiBP) | Baseline; Week One; Two Week (End of Study)
  The survey contains six items three items measure depressive symptoms (depressed mood, fidgeting, and fatigue), two items measure manic symptoms (increased energy, rapid speech), and one item measures both (irritability). Participants rate symptoms on an ordinal scale: 0 = absent/normal, 1 = mild, 2 = moderate, 3 = severe. Items can be aggregated into two scores to reflect depressive symptom severity and manic symptom severity. Higher depression and manic scores reflect more severe depressive and manic symptoms, respectively. Since item responses range from 0 to 3, the depression score ranges from 0 (no symptoms) to 21 (all depressive symptoms are severe), whereas the manic score ranges from 0 (no symptoms) to 15 (all manic symptoms are severe).
Change in Altman Self-Rating Mania Scale - 5-Item Self Rating Mania Scale (ASRM) | Baseline; Week One; Two Week (End of Study)
  The Altman Self-Rating Mania Scale is a 5-item self-rating mania scale designed to assess the presence and/or severity of manic symptoms. Each item on the measure is rated on a 5-point scale (i.e., 1 to 5) with the response categories having different anchors depending on the item. The Altman Self-Rating Mania Scale score range from 5 to 25 with higher scores indicating greater severity of manic symptoms.
Change in the Hamilton Depression Rating Scale - 21-Item for the Assessment of Depression Severity (HAM-D) | Baseline; Day 1-2; Day 3-5; Week One; Day 9-10; Day 11-12; Week Two (End of Study)
  The scale is widely available and has two common versions with either 1 and is scored between 0 and 4 points. Scoring is based on the 17-item scale and scores of 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression; the maximum score being 52 on the 17-point scale.
Change in the Patient Health Questionnaire - 9-Item Measuring the Severity of Depression Symptoms (PHQ-9) | Baseline; Week One; Two Week (End of Study)
  Self-reported measurement of the severity of depression symptoms experienced within the last two weeks. The survey consists of 9 items. Participants are asked to rate each symptom of depression on a Likert scale, providing a score between 0 (not at all) and 3 (nearly every day). This yields a total score ranging from 0 (minimal depression) to 27 (severe depression). Higher scores thus indicate a greater severity of depressive symptoms, and are interpreted in the following manner: a score of 0-4 indicates minimal depression, a score of 5-9 indicates mild depression, a score of 10-14 indicates moderate depression, a score of 15-19 indicates moderately severe depression, and a score of 20-27 indicates severe depression.
Change in the General Anxiety Disorder Questionnaire- 7-Item Measuring Severity of Anxiety Symptoms (GAD-7) | Baseline; Week One; Two Week (End of Study)
  Self-reported measurement of the severity of anxiety symptoms experienced within the last two weeks. It consists of 7 scored items and one follow-up question. Each of the 7 scored items generates a value from 0 (not at all) to 3 (nearly every day), yielding a total score ranging from 0 to 21, with higher scores indicating more severe symptoms of anxiety. These scores are interpreted in the following manner: a score of 0-4 indicates little or no anxiety, a score of 5-9 indicates mild anxiety, a score of 10-14 indicates moderate anxiety, and a score of 15-21 indicates severe anxiety. Generally, a score of 10 or above is considered to be a clinical cutoff implying that the respondent may be suffering from a general anxiety disorder.
Change in The Morning Evening Questionnaire - 19-Item Self-Assessment Questionnaire for Sleep Rhythms, Habits and Fatigue (MEQ) | Baseline; Week One; Two Week (End of Study)
  This questionnaire has 19 questions, each with a number of points. Scores can range from 16-86. Scores of 41 and below indicate "evening types." Scores of 59 and above indicate "morning types." Scores between 42-58 indicate "intermediate types."
Change in The Pittsburgh Sleep Quality Index - 18-Item Self-Assessment to Evaluate Sleep Quality (PSQI) | Baseline; Week One; Two Week (End of Study)
  The Pittsburg Sleep Quality Index Questionnaire is self-administered questionnaire designed to evaluate sleep quality consisting of 18 items that in turn are comprised of seven components, which include subjective sleep quality, sleep duration, sleep onset, habitual sleep efficiency, sleep disturbances, use of sleeping medications and daytime dysfunction. Each weighted equally on a 0-3 scale to be summed to yield a global PSQI score, which ranges between 0 and 21, where the higher the scores, the worse the sleep quality. The investigators will only be using questions 1-4 and 6.
Change in The Leeds Sleep Evaluation Questionnaire - 10-Item Self-Rating Scale of Sleep Behavior (LEEDS) | Baseline; Week One; Two Week (End of Study)
  The Leeds Sleep Evaluation Questionnaire comprises ten self-rating 100-mm-line analogue questions concerned with aspects of sleep and early morning behavior. A 10-cm line separates the two halves of each question. The questionnaire instructions are" "Each question is answered by placing a vertical mark on the answer line. If no change was experienced then place your mark in the middle of the line. If a change was experienced then the position of your mark will indicate the nature and extent of the change, i.e. large charges near the ends of the line, small changes near the middle." The questionnaire monitors subjectively perceived changes in sleep. Improvements in the self-reported ratings relate to improved perceived quality of sleep.
Change in the Pre-Sleep Arousal Scale - 16-Item Self-Rated Scale of Symptoms of Arousal at Bedtime (PSAS) | Baseline; Week One; Two Week (End of Study)
  The Pre-Sleep Arousal Scale contains 16 items, each rated on a 5-point scale that describes symptoms of arousal at bedtime. Eight items evaluates cognitive arousal and eight evaluates somatic arousal. Total score scores range from 16 to 80, with higher scores suggest higher pre-sleep arousal.
Change Circadian Rhythms | Inferred from melatonin/cortisol curves, rest-activity cycle (wrist actigraphy), heart rate/temperature monitoring, Electroencephalography
  Substudy for subsample (measured at Baseline and Week One)

CONTACTS AND LOCATIONS:
Overall Officials: Jess G Fiedorowicz, MD, PhD, Principal Investigator — Head and Chief, Department of Mental Health, The Ottawa Hospital
Locations (2):
- Canada (2):
  - Ottawa Hospital Research Insitute, Ottawa, Ontario
  - L'Hôpital Montfort, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data to other researchers.

REFERENCES:
- [Derived] Fiedorowicz JG, Mikhail E, Solmi M, Burns JK, Yu J, Siddiqi S, Nguyen T, Smith AL, Robillard R; Ottawa Sunglasses at Night Investigators and Coordinators. The Ottawa sunglasses at night study: A randomized controlled trial of blue-blocking glasses for mania. J Affect Disord. 2026 Apr 1;398:120910. doi: 10.1016/j.jad.2025.120910. Epub 2025 Dec 18. PMID 41421618